CLINICAL TRIAL: NCT02932306
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Vehicle- Controlled, 2-Arm, Parallel Group Comparison Study Comparing the Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Brief Title: Efficacy and Safety of IDP-121 and IDP-121 Vehicle Lotion in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-121A-301
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-121 Lotion (Experimental): IDP-121 lotion (tretinoin 0.05 percent [%]) will be applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
  Interventions: Drug: IDP-121 Lotion
- IDP-121 Vehicle Lotion (Placebo Comparator): IDP-121 lotion vehicle will be applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
  Interventions: Drug: IDP-121 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-121 Lotion — IDP-121 lotion will be applied as per the instructions provided by the investigational center staff.
  Arms: IDP-121 Lotion
Drug: IDP-121 Vehicle Lotion — IDP-121 vehicle lotion will be applied as per the instructions provided by the investigational center staff.
  Arms: IDP-121 Vehicle Lotion

SUMMARY:
The objective of this study was to evaluate the efficacy, safety, and tolerability of a once daily topical application of IDP-121 Lotion compared with its vehicle (IDP-121 Vehicle Lotion) in participants with moderate to severe acne vulgaris (acne) (that is, acne having an Evaluator's Global Severity Score [EGSS] of 3 [moderate] or 4 [severe]).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 9 years of age and older.
* Written and verbal informed consent must be obtained. Participants less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if participant reaches age of consent during the study they should be re-consented at the next study visit).
* Participant must have a score of 3 (moderate) or 4 (severe) on the EGSS assessment at the screening and baseline visit

Key Exclusion Criteria:

* Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gram-negative folliculitis.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Participants with a facial beard or mustache that could interfere with the study assessments.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Theisen, Study Chair — TKL Research, Inc.
Locations (39):
- United States (39):
  - Valeant Site 36, Guntersville, Alabama
  - Valeant Site 14, Phoenix, Arizona
  - Valeant Site 28, Hot Springs, Arkansas
  - Valeant Site 38, Fountain Valley, California
  - Valeant Site 34, Manhattan Beach, California
  - Valeant Site 23, Oceanside, California
  - Valeant Site 35, Rancho Cucamonga, California
  - Valeant Site 20, San Diego, California
  - Valeant Site 32, Denver, Colorado
  - Valeant Site 10, Shelton, Connecticut
  - Valeant Site 02, Boynton Beach, Florida
  - Valeant Site 15, Coral Gables, Florida
  - Valeant Site 37, Miami, Florida
  - Valeant Site 39, Pembroke Pines, Florida
  - Valeant Site 01, West Palm Beach, Florida
  - Valeant Site 19, Boise, Idaho
  - Valeant Site 04, Arlington Heights, Illinois
  - Valeant Site 27, Carmel, Indiana
  - Valeant 12, Plainfield, Indiana
  - Valeant Site 09, Louisville, Kentucky
  - Valeant Site 16, Louisville, Kentucky
  - Valeant Site 33, Needham, Massachusetts
  - Valeant Site 11, Warren, Michigan
  - Valeant Site 08, Omaha, Nebraska
  - Valeant Site 25, Omaha, Nebraska
  - Valeant Site 13, Berlin, New Jersey
  - Valeant Site 03, Albuquerque, New Mexico
  - Valeant Site 26, New York, New York
  - Valeant Site 31, Stony Brook, New York
  - Valeant 05, Gresham, Oregon
  - Valeant Site 22, Fort Washington, Pennsylvania
  - Valeant Site 24, Charleston, South Carolina
  - Valeant Site 06, Dallas, Texas
  - Valeant Site 30, Houston, Texas
  - Valeant Site 17, Pflugerville, Texas
  - Valeant Site 07, San Antonio, Texas
  - Valeant 18, Webster, Texas
  - Valeant Site 29, Salt Lake City, Utah
  - Valeant Site 21, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tyring SK, Kircik L, Pariser DM, Woolery-Lloyd HC, Harper JC, Bhatt V, Pillai R, Guenin E. The Effects of Once-Daily Tretinoin 0.05% Lotion on Quality of Life in Patients with Moderate-to-Severe Acne Vulgaris. Am J Clin Dermatol. 2020 Dec;21(6):891-899. doi: 10.1007/s40257-020-00559-3. PMID 32886337

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either IDP-121(tretinoin 0.05 percent [%]) Lotion or IDP-121 Vehicle Lotion.
Groups:
- IDP-121 Lotion: IDP-121 lotion (tretinoin 0.05%) was applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
- IDP-121 Vehicle Lotion: IDP-121 lotion vehicle was applied topically to the face of participants with moderate to severe acne, once daily for 12 weeks.
Period: Overall Study
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Started | 406 | 414
Intent-to-treat (ITT) Population (All randomized participants who received study drug.) | 406 | 414
Safety Population (All randomized participants with ≥1 confirmed dose of study drug and ≥1 post baseline evaluation.) | 378 | 385
Completed | 338 | 337
Not Completed | 68 | 77
Not completed — Withdrawal by Subject | 16 | 25
Not completed — Adverse Event | 3 | 0
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Noncompliance with Study Drug | 1 | 1
Not completed — Lost to Follow-up | 36 | 40
Not completed — Withdrawal by Parent or Guardian | 6 | 8
Not completed — Lack of Efficacy | 0 | 2
Not completed — Worsening condition | 2 | 0
Not completed — Withdrew due to burning,itching,stinging | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion | Total
Number analyzed (Participants) | 406 | 414 | 820
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (7.15) | 20.5 (7.26) | 20.4 (7.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 247 | 476
  Male | 177 | 167 | 344
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 146 | 168 | 314
  Not Hispanic or Latino | 260 | 246 | 506
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 3 | 5 | 8
  Black or African American | 75 | 72 | 147
  White | 296 | 308 | 604
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Evaluator's Global Severity Score (EGSS) [Count of Participants; unit: Participants] — EGSS was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. Population: 'Number analyzed' signifies participants evaluable for this parameter.
  Participants
    0 - Clear: number analyzed (Participants) | 405 | 414 | 819
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear: number analyzed (Participants) | 405 | 414 | 819
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild: number analyzed (Participants) | 405 | 414 | 819
    2 - Mild | 0 | 0 | 0
    3 - Moderate: number analyzed (Participants) | 405 | 414 | 819
    3 - Moderate | 368 | 366 | 734
    4 - Severe: number analyzed (Participants) | 405 | 414 | 819
    4 - Severe | 37 | 48 | 85
Noninflammatory Lesion Count [Mean (Standard Deviation); unit: lesion count] | 38.0 (15.67) | 39.2 (16.70) | 38.6 (16.20)
Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesion count] | 26.1 (5.56) | 26.4 (5.63) | 26.3 (5.60)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Mean Noninflammatory Lesion Count to Week 12
Description: Noninflammatory lesions were defined as follows: Open comedones (blackhead) - plugged hair follicle with dilated/open orifice, black in color; and Closed comedones (whitehead) - plugged hair follicle: small opening at skin surface. For noninflammatory facial lesions, open and closed comedones were recorded as a single count.
Time Frame: Baseline (Day 0), Week 12
Population: ITT population included all randomized participants who received study drug. Multiple imputation (Markov Chain Monte Carlo [MCMC]) was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: lesion count
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 406 | 414
lesion count | -17.8 (15.18) | -10.6 (16.07)
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using analysis of covariance (ANCOVA) with factors of treatment group and analysis center and the respective baseline lesion count as a covariate; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05

2. Primary Outcome: Absolute Change From Baseline in Mean Inflammatory Lesion Count to Week 12
Description: Inflammatory lesions were defined as follows: Papule - a solid, elevated lesion less than 5 millimeters (mm); and Pustule - an elevated lesion containing pus less than 5 mm. For inflammatory facial lesions, papules and pustules were recorded as a single count, while nodular lesions were counted and recorded separately.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants who received study drug. Multiple imputation (MCMC) was used to impute missing values.
Measure: Least Squares Mean (Standard Deviation); unit: lesion count
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 406 | 414
lesion count | -13.1 (10.50) | -10.2 (10.87)
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using ANCOVA with factors of treatment group and analysis center and the respective baseline lesion count as a covariate; Test type: Superiority; p < 0.001, ANCOVA — Threshold for significance at 0.05

3. Primary Outcome: Percentage of Participants With Treatment Success at Week 12
Description: Treatment success was defined as at least a 2-grade reduction from Baseline in EGSS score and an EGSS score equating to "Clear" or "Almost Clear". EGSS was based on a 5-point scale ranging from 0 to 4; where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants who received study drug and evaluable for EGSS score. Multiple imputation (MCMC) was used to impute missing values. 1 participant was excluded from analysis of dichotomized EGSS because EGSS was not performed at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 405 | 414
percentage of participants | 16.5 | 6.9
Statistical Analysis 1: Comparison: IDP-121 Lotion vs IDP-121 Vehicle Lotion; Analysis was performed using a logistic regression test (using Firth's Penalized Likelihood) with factors of treatment group and analysis center; Test type: Superiority; p < 0.001, Regression, Logistic — Threshold for significance at 0.05

4. Secondary Outcome: Percent Change From Baseline in Noninflammatory Lesion Count to Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 406 | 414
percent change | -47.5 (41.92) | -27.3 (43.96)

5. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count to Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
Number analyzed (Participants) | 406 | 414
percent change | -50.9 (40.72) | -40.4 (42.29)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to Week 12
Description: Safety population included all randomized participants who were presumed to have used study drug at least once and who provided at least 1 post baseline evaluation.
Arm/Group | IDP-121 Lotion | IDP-121 Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/378 | 0/385
Serious Adverse Events (participants affected / at risk) | 5/378 | 2/385
Other Adverse Events (participants affected / at risk) | 0/378 | 0/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | IDP-121 Lotion (N=378) | IDP-121 Vehicle Lotion (N=385)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2/229 | 1/247 — This is a gender-specific AE. Only female participants were at risk.
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/229 | 1/247 — This is a gender-specific AE. Only female participants were at risk.
Appendicitis (Infections and infestations) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT02932306/Prot_SAP_000.pdf